CLINICAL TRIAL: NCT03906799
Title: A Placebo-controlled, Double-blind, Randomized, Dose-finding Phase II Study on OMT-28 in MaIntenance of Sinus Rhythm After Electrical Cardioversion in Patients With Persistent Atrial Fibrillation (PROMISE-AF)
Brief Title: Study on OMT-28 in Maintenance of Sinus Rhythm in Patients With Persistent Atrial Fibrillation (AF)
Acronym: PROMISE-AF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Omeicos Therapeutics GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OMT28-C0201
Record Dates: First submitted 2019-03-20; First posted 2019-04-08 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2019-03

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; Electrical Cardioversion; Dose-finding
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Low OMT-28 (Experimental): Verum, low OMT-28
  Interventions: Drug: OMT-28
- Middle OMT-28 (Experimental): Verum, middle OMT-28
  Interventions: Drug: OMT-28
- High OMT-28 (Experimental): Verum, high OMT-28
  Interventions: Drug: OMT-28
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: OMT-28 — 1 capsule given daily orally from Visit 3 (Day 1) to Visit 8 (Day 99 ± 3 days).
  Arms: High OMT-28; Low OMT-28; Middle OMT-28
Drug: Placebo — 1 capsule given daily orally from Visit 3 (Day 1) to Visit 8 (Day 99 ± 3 days).
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, dose-finding, placebo-controlled, parallel group, multicenter, phase II study to evaluate the efficacy, safety, and popPK of three different doses of OMT-28 given once daily versus placebo in patients with persistent AF.

DETAILED DESCRIPTION:
This is a randomized, double-blind, dose-finding, placebo-controlled, parallel group, multicenter, phase II study to evaluate the efficacy, safety, and popPK of three different doses of OMT-28 given once daily versus placebo in patients with persistent AF. At randomization, the duration of the current episode of persistent AF must be shown to be greater than 7 days and not greater than 3 months, as confirmed by two ECGs (one ECG must be a 12-lead ECG) and further patient enquiry (including doctor visits, hospital admissions, symptom onset, etc.).

A sample size re-evaluation will be performed to avoid an underpowered study because of imprecise estimates for the study population or overoptimistic parameter estimates. Therefore, an interim analysis will re-evaluate sample size assumptions after approximately 15 patients per study arm (~50 % of planned sample) have completed the treatment phase (Visit 8) of the study. Predefined rules will govern the decision for adjustment of sample size.

Patients will be monitored for cardiac events throughout the study using an Implantable Cardiac Monitor (ICM). Safety will be monitored throughout the study. Blood samples will be collected in pre-specified windows for popPK analysis and at pre-specified timepoints for PK/PD analysis. Patients will be provided with a diary to record timing of drug administration and clinical symptoms while not on site. Diaries will be reviewed and checked for compliance at each non-resident visit to the clinical site.

ELIGIBILITY:
Inclusion Criteria:

* Males or females between 18 and 85 years of age.
* Patients with persistent AF for > 7 days but ≤ 3 months suitable for electrical DCC.
* Male patients must be surgically sterile for at least 90 days or will be required to use a male condom with spermicide, and will refrain from donating sperm from the time of the first dose until 90 days after the last dose of study medication.
* Females of childbearing potential (postmenarchal, not surgically sterile, premenopausal) will agree to follow contraception requirements from the time of signing the Informed Consent Form (ICF) until 90 days after the last administration of study drug.
* Willing and able to give written informed consent before any study-related procedure.
* Willing and able to attend all the visits scheduled in the study.

Main Exclusion Criteria:

* Patients with known concurrent temporary secondary causes of AF
* Patients that have undergone surgical or catheter ablation for AF or atrial flutter.
* Patients with an existing cardiac treatment device, pacemaker, implantable cardioverter defibrillator, or cardiac resynchronization therapy.
* Patients with a history of ECG abnormalities that, in the opinion of the investigator (or designee), render the patient unsuitable for the study.
* Patients with congestive heart failure (NYHA class III and IV).
* Patients with left atrium size ≥ 55 mm.
* Patients with left ventricular ejection fraction ≤ 40 %.
* Known presence of a thrombus in the left atrial appendage, left atrium, left ventricle, aorta, or intracardial mass.
* Patients with moderate or severe mitral stenosis, mitral valve rheumatic disease, unresected atrial myxoma, or a mechanical heart valve and/or other conditions, such as pulmonary embolism, considered to be formal indication for conventional anticoagulation.
* Patients with any acute coronary event, stroke, or percutaneous coronary intervention within 6 months prior to randomization or who are receiving dual antiplatelet therapy.
* Uncontrolled/therapy-resistant bradycardia and/or uncontrolled/therapy-resistant hypertension within a 3-month period prior to randomization.
* Patients having more than two DCCs in the last 6 months. Any unsuccessful pharmacological and/or electrical cardioversion (within prior 3 months).
* Patients with signs of bleeding or conditions associated with a high risk of bleeding.
* Patients taking antiarrhythmic agents within 3 days of planned randomization will be excluded.
* Patients concurrently participating in another study or unable to communicate.
* Patients with active cancer, chronic kidney disease or intercurrent illness.
* Pregnant or breastfeeding women.
* Patients taking concomitant medication.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2019-03-19 (Actual); Primary Completion 2019-11-20 (Actual); Study Completion 2020-03-20 (Actual)

PRIMARY OUTCOMES:
Assessment of AF Burden After OMT-28 Administration | Up to 4.5 months
  To assess the AF burden, based on data collected via the implantable cardiac monitor BioMonitor 2-AF, of three different doses of OMT-28 administered once daily versus placebo in the maintenance of normal sinus rhythm after electrical direct current cardioversion (DCC) in patients with persistent AF

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | Up to 4.5 months
  To assess the incidence of treatment-emergent Adverse Events of three different doses of OMT-28 administered once daily versus placebo after electrical DCC in patients with persistent AF.
Assessment of Pharmacokinetic (PK) Parameters of OMT-28 - AUC | Up to 3.5 months
  To assess the pharmacokinetic (PK) parameter AUC of OMT-28 administered once daily in patients with persistent AF, by means of population PK (popPK) analysis.
Assessment of Pharmacokinetic (PK) Parameters of OMT-28 - Cmax | Up to 3.5 months
  To assess the pharmacokinetic (PK) parameter Cmax of OMT-28 administered once daily in patients with persistent AF, by means of population PK (popPK) analysis.

OTHER OUTCOMES:
Concentration of NT-proBNP | Up to 3.5 months
  To assess the concentration of the exploratory, pharmacodynamic (PD) parameter NT-proBNP after once-daily administration of OMT-28 or placebo in patients with persistent AF.
Concentration of GDF-15 | Up to 3.5 months
  To assess the concentration of the exploratory, pharmacodynamic (PD) parameter GDF-15 after once-daily administration of OMT-28 or placebo in patients with persistent AF.
Concentration of MMP-9 | Up to 3.5 months
  To assess the concentration of the exploratory, pharmacodynamic (PD) parameter MMP-9 after once-daily administration of OMT-28 or placebo in patients with persistent AF.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Gebauer, Dr.med., Study Director — Managing Director
Locations (25):
- Bulgaria (3):
  - Site 401, Sofia
  - Site 404, Stara Zagora
  - Site 402, Varna
- Czechia (3):
  - Site 301, Kolín
  - Site 303, Pilsen
  - Site 302, Slaný
- Hungary (6):
  - Site 205, Budapest
  - Site 201, Budapest
  - Site 203, Debrecen
  - Site 206, Hódmezővásárhely
  - Site 202, Pécs
  - Site 204, Zalaegerszeg
- Ukraine (13):
  - Site 102, Cherkasy
  - Site 110, Ivano-Frankivsk
  - Site 104, Kharkiv
  - Site 107, Kharkiv
  - Site 108, Khmelnytskyi
  - Site 113, Kiev
  - Site 106, Kiev
  - Site 101, Kiev
  - Site 109, Kiev
  - Site 112, Kiev
  - Site 105, Odesa
  - Site 103, Uzhhorod
  - Site 111, Zhytomyr

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schunck WH, Konkel A, Fischer R, Weylandt KH. Therapeutic potential of omega-3 fatty acid-derived epoxyeicosanoids in cardiovascular and inflammatory diseases. Pharmacol Ther. 2018 Mar;183:177-204. doi: 10.1016/j.pharmthera.2017.10.016. Epub 2017 Nov 7. PMID 29080699
- [Background] Fischer R, Konkel A, Mehling H, Blossey K, Gapelyuk A, Wessel N, von Schacky C, Dechend R, Muller DN, Rothe M, Luft FC, Weylandt K, Schunck WH. Dietary omega-3 fatty acids modulate the eicosanoid profile in man primarily via the CYP-epoxygenase pathway. J Lipid Res. 2014 Jun;55(6):1150-64. doi: 10.1194/jlr.M047357. Epub 2014 Mar 16. PMID 24634501
- See also: OMEICOS Therapeutics GmbH — http://www.omeicos.com/